CLINICAL TRIAL: NCT06927479
Title: The Effect of the Electronic Decision Support System Developed for the Use of Informal Caregivers on Preventing the Risk of Pressure Sore and Urinary Infection in Patients Receiving Home Care
Brief Title: The Effect of an Electronic Decision Support System on Preventing Pressure Ulcers and Urinary Infectionsin Home Care
Acronym: e-CARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sebahat Gozum, Prof.Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TBAEK-257
Record Dates: First submitted 2025-03-20; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Support of the Family as a Caregiving System
Keywords: decision support system; pressure ulcer; urinary infection; home care; infection risk; dependent patients; informal caregiver
MeSH Terms: conditions — Pressure Ulcer; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Caregivers in this group will use the electronic decision support system (E-DSS) provided via a mobile-compatible web page. E-DSS will be used to optimize the daily care management of patients and to reduce the risk of pressure ulcers and the risks that predict this risk, such as nutrition and hydration, position changes and in-bed activities. E-DSS will analyze the data obtained from the participants and provide personalized recommendations. Caregivers in the intervention group will receive this training over a period of two weeks, with ongoing support and reinforcement provided throughout the eight-week intervention period via the Electronic Decision Support System (E-DSS).
  Interventions: Other: Training about Electronic Decision Support System
- Control group (No Intervention): This group will contiue with home care services by Health Ministriy ot Turkiye

INTERVENTIONS:
Other: Training about Electronic Decision Support System — 1. System Registration and Usage
  2. Pressure Ulcer Prevention
  3. Urinary Infection Prevention
  4. Nutrition and Hydration Management
  5. Physical Activity and In-Bed Mobilization
  6. Emergency Management and Reporting
  7. Continuous Monitoring and Feedback
  Arms: Intervention group

SUMMARY:
The home care of fully dependent patients is often provided by informal family caregivers. Therefore, caregivers need support systems to make the right decisions during home care to prevent pressure ulcers and urinary infections. This study aims to evaluate the impact of using an electronic decision support system (E-DSS), offered through a mobile-compatible webpage, on preventing the risk of pressure ulcers and urinary infections in fully dependent patients receiving home healthcare services.

The study is planned in two phases. In the first phase, the development of the electronic decision support system to be provided through a mobile-compatible webpage is targeted. In the second phase, a randomized controlled trial will be conducted to assess the usability of the developed decision support system by caregivers.

For the project, patients with a Barthel Index score between 0-20 (if an insufficient number of patients is available, those scoring between 21-61 will also be included) will be selected and divided into intervention and control groups. Caregivers of the intervention group will use the electronic decision support system via a mobile-compatible webpage for eight weeks to receive guidance on preventing pressure ulcers, urinary infection prevention strategies, in-bed mobilization, and nutrition recommendations. Caregivers in the control group will continue with the routine practices of the home healthcare services provided by the Turkish Ministry of Health.

The study outcomes will be evaluated at the beginning and at the ninth week using the Braden Pressure Ulcer Risk Scale, the Ghent Global IAD Classification Tool (GLOBIAD), the ISTAP Skin Tear Classification System, urinalysis (UA), the Urine Color Scale, and the Mini Nutritional Assessment-Short Form (MNA-SF). Additionally, at the end of the study, caregivers in the intervention group will be assessed using the System Usability Scale (SUS-TR), the Mobile Application Usability Scale, the Mobile Application Loyalty Scale, and the Mobile Application Willingness to Use Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving home healthcare services.
2. Patients with a total Barthel Index score of 0-20 (fully dependent) and 21-61 (severely dependent).
3. Caregivers who are familiar with using mobile devices and voluntarily agree to participate.

Exclusion Criteria:

1. Patients with a Barthel Index score of 62 or above.
2. Patients with an acute medical condition (e.g., hospitalization due to infection or newly developed severe illness).
3. Caregivers with cognitive or technological limitations preventing
4. Caregivers who are not literate in Turkish and unable to use the application.
5. Terminal-stage patients* with a life expectancy of a short period.
6. Caregivers with severe cognitive impairment (e.g., advanced-stage dementia) or untreated psychiatric disorders (e.g., schizophrenia).
7. Patients without an informal caregiver providing care at home.
8. Patients with an existing urinary infection based on hospital urinalysis records.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Prevention of Pressure Ulcer Risk | Baseline, 5th and 9th weeks
  Change in pressure ulcer risk scores measured by the Braden Pressure Ulcer Risk Scale

SECONDARY OUTCOMES:
Nutritional and Hydration Status | Baseline, 5th and 9th weeks
  This change will be evaluate by Mini Nutritional Assesment Short Form
Prevention of Urinary Infection Risk | Baseline, 5th and 9th weeks.
  Change in urinary infection risk based on urinalysis (UA) results

IPD SHARING:
Plan to Share IPD: Undecided
This is a continuing doctorate thesis. We will share ID when our thesis finished.